CLINICAL TRIAL: NCT05368662
Title: Quality of Life and Quality of Sleep Studies in Children with Home Care Ventilation in Two Regions of France Pays De Loire and Bretagne
Brief Title: Quality of Life and Quality of Sleep Studies in Children with Home Care Ventilation in the West of France
Acronym: EQuaViSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 49RC20_0239
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Quality of Life; Non Invasive Ventilation
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with home ventilation (Experimental)
  Interventions: Other: Quality of life and sleep questionnaire

INTERVENTIONS:
Other: Quality of life and sleep questionnaire — Evaluation of quality of life and quality of sleep by questionnaires

SUMMARY:
Home ventilation in children, invasive or non invasiv,e is an interesting treatment for different disease which cause chronic respiratory impairement. The aim of this treatment is to support alveolar hypoventilation. Concerned diseases are : neuro-muscular disease, upper airways pathologies, whest wall or lung pathologies, central control ventilation disease. Prevalence of home children ventilation is in augmentation in France. The last national study in 2021 about infants show a prevalence of 9.3/100 000. Advantages with home children ventilation in addition of improvement of survey, it can observe improvement of quality of life and improvement of the quality of their sleep. Quality of life is a thematic less studying. Last studies show an impairment of quality of life in all thematics compare to children with no disease but also with infants whith chronic diseases. This study were about few numbers of patients. The aim of this study is to evaluate the quality of life and the quality of sleep in children with home ventilation to complete the actual littérature to improve the respiratory care of this population.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 6 months to 17 years treated with non-invasive ventilation at home for at least 1 month
* Follow-up in one of the five centers participating in the study (Angers, Nantes, Le Mans, Rennes and Brest)
* Informed consent form signed by both parents, or holder of parental authority, for the participation of their child
* To be affiliated or beneficiary of social security

Exclusion Criteria:

* Parents with poor command of the French language, implying not being able to complete the various questionnaires
* Refusal of the child to participate in the study

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2022-11-11 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-09-24 (Estimated)

PRIMARY OUTCOMES:
Quality of life in children with home care ventilation | 30 months
  The quality of life of this population is assessed using the generic PedsQL 4.0 score. The questions are classified according to different categories regardless of age: physical capacity, emotional functioning, social relationships and schooling, or for children under 2 years old, relationship life and cognitive functioning. The evaluation relates to the past month. The questionnaire presents different questions depending on the age group

CONTACTS AND LOCATIONS:
Locations (1):
- CHU, Angers, Maine et Loire, France

IPD SHARING:
Plan to Share IPD: No